CLINICAL TRIAL: NCT03652337
Title: Meibomian Gland Dysfunction Management to Relieve Contact Lens Discomfort
Brief Title: Meibomian Gland Dysfunction Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Collaborators: American Academy of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-04-003
Record Dates: First submitted 2018-06-19; First posted 2018-08-29 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Contact Lens Discomfort; Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BlephEx (Experimental): The subjects who are enrolled in this arm will undergo electronic lid margin debridement using the BlephEx instrument.
  Interventions: Device: BlephEx
- Manual debridement (Experimental): The subjects who are enrolled in this arm will undergo manual lid margin debridement using a stainless steel ophthalmic golf spud.
  Interventions: Device: Manual debridement

INTERVENTIONS:
Device: BlephEx — Electronic lid margin debridement
  Arms: BlephEx
Device: Manual debridement — Manual lid margin debridement
  Arms: Manual debridement

SUMMARY:
The purpose of this study is to compare electronic debridement of the eyelid margin (BlephEx) to manual debridement of the eyelid margin as treatment options for patients intolerant to contact lens wear consequent to Meibomian gland dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Habitual contact lens wearers whose contact lens wear time has reduced due to MGD will be preferentially considered for this study. Subjects who currently cannot wear contact lenses due to MGD may be considered on a case-by-case basis.

Exclusion Criteria:

* Subjects who are currently using any prescription ophthalmic medications (such as antibiotics, steroids and immunomodulatory drugs) will be excluded from participation.
* Subjects who have active ocular infections will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Symptomatic relief | 60 days
  Betterment of symptoms (improvement in contact lens discomfort) will be measured using two different surveys - Ocular Surface Disease Index (OSID) and Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8). The OSDI scores can range from 0 to 100. The CLDEQ-8 scores can range from 0 to 37. In both the questionnaires, a lowering of the score during follow-up visits represents a betterment of symptoms suffered by the patient. The numerical change in the scores on these two questionnaires will be documented as the change in symptom profile of the patient (betterment / worsening / stability).

SECONDARY OUTCOMES:
Meibography | 60 days
  Meibomian gland imaging will be performed to document any changes in the Meibomian gland during the study period.
Lissamine green staining grade of the lid margin | 60 days
  The lid margin will be stained with Lissamine green dye. For the purpose of this study, Lissamine green staining of the eyelid margins will be graded from 0 to 4. (Zero representing "normal" or "no" staining; Four representing the highest degree of staining). During the course of the study, a decrease in lid margin staining will indicate a betterment of the health of the eyelid margin.
Inflammatory activity | 60 days
  The presence or absence of Matrix Metalloproteinase-9 (MMP-9) in the tear fluid will be documented during the study visits. Presence of MMP-9 in the tear fluid indicates the presence of inflammatory activity in the tear fluid.
Tear break-up time | 60 days
  Improvement in non-invasive tear break-up time measurement will be an objective outcome of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Srihari Narayanan, OD, PhD, Principal Investigator — Professor
Locations (1):
- Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Result] Korb DR, Blackie CA. Debridement-scaling: a new procedure that increases Meibomian gland function and reduces dry eye symptoms. Cornea. 2013 Dec;32(12):1554-7. doi: 10.1097/ICO.0b013e3182a73843. PMID 24145633